CLINICAL TRIAL: NCT06327035
Title: Neurological Recovery of the Paretic Lower Limb and Balance and Walking Abilities in the Subacute Phase of Stroke in Patients Hospitalized in Medical and Rehabilitation Units: A Prospective Multicenter Longitudinal Study
Brief Title: Evolution of Walking Abilities in Subacute Stroke Patients Hospitalized in Neurorehabilitation Center
Acronym: PROWALK
Status: Recruiting | Type: Observational
Sponsor: Clinique Les Trois Soleils (Other)
Collaborators: Le Normandy (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2023-A02660-45
Record Dates: First submitted 2024-03-15; First posted 2024-03-25 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-03

CONDITIONS: Stroke; Gait, Hemiplegic
Keywords: stroke; lower limb; gait recovery; balance
MeSH Terms: conditions — Stroke; Gait Disorders, Neurologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Gait rehabilitation — Assessment of gait and balance abilities after stroke during neurorehabilitation from the subacute phase of stroke to 6 months after stroke.
  The assessments will be carried out on entrance to the neurological center, then at 1 ,3 and 6 months and on hospital discharge.

SUMMARY:
The goal of this observational study is to describe the evolution of gait recovery during the subacute phase of stroke up to six months after stroke, in patients hospitalized in medical and neurological rehabilitation units.

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalized in one of the investigating centers after acute/subacute stroke.
* Affiliated to a social security scheme

Exclusion Criteria:

* Opposed to its participation in this study
* Neurodegenerative disease impacting gait prior to stroke onset
* Patient not walking before stroke
* Progressive pathology with life-threatening consequences within 6 months
* Patient under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke patient hospitalized in one of the investigating centers during acute/subacute phase.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-03-26 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Functional Ambulation Classification | Functional Ambulation Classification will be carried out within 72 hours of admission to the neurological center, then at 1, 3 and 6 months, and at discharge from hospital (assessed up to 5 days).
  The Functional Ambulation Categories (FAC) is a 6-point functional walking test that evaluates ambulation ability.

SECONDARY OUTCOMES:
Postural Assesment Scale for Stroke Patient | Postural Assesment Scale for Stroke Patient will be carried out within 72 hours of admission to the neurological center, then at 1, 3 and 6 months, and at discharge from hospital (assessed up to 5 days).
  The Postural Assessment Scale for Stroke Patients (PASS) assesses balance in lying, sitting and standing positions. It was designed specifically for patients with stroke and is suitable for all individuals regardless of postural performance.
  The PASS consists of a 4-point scale where items are scored from 0 - 3. The total score ranges from 0 - 36, the higher the score is, the more favourable the balance in stroke patients.
Timed Up and Go | Timed Up and Go will be carried out within 72 hours of admission to the neurological center, then at 1, 3 and 6 months, and at discharge from hospital (assessed up to 5 days).
  The Timed Up and Go is a general physical performance test used to assess mobility, balance and locomotor performance. More specifically, it assesses the ability to perform sequential motor tasks relative to walking and turning.
10-Meter Walk Test | 10-Meter Walk Test will be carried out within 72 hours of admission to the neurological center, then at 1, 3 and 6 months, and at discharge from hospital (assessed up to 5 days).
  The 10 Metre Walk Test is a performance measure used to assess walking speed in meters per second over a short distance
6Minute-Walk Test | 6Minute-Walk Test will be carried out within 72 hours of admission to the neurological center, then at 1, 3 and 6 months, and at discharge from hospital (assessed up to 5 days).
  The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
Motricity Index | Motricity Index will be carried out within 72 hours of admission to the neurological center, then at 1, 3 and 6 months, and at discharge from hospital (assessed up to 5 days).
  The Motricity Index (MI) is an ordinal method of measuring limb strength. The total score ranges from 0 - 100, with the higher numbers representing good muscle strength.

CONTACTS AND LOCATIONS:
Overall Officials: Christophe T Duret, MD, Principal Investigator — Les Trois Soleils
Locations (3):
- France (3):
  - Le Normandy, Granville, Normandy
  - Clinique Les Trois Soleils, Boissise-le-Roi
  - La Clinique Les Trois Soleils, Boissise-le-Roi

IPD SHARING:
Plan to Share IPD: Undecided